CLINICAL TRIAL: NCT06637657
Title: Guided Optimisation of Long-term Disease rEduction in secoNdary Prevention of CVD (GOLDEN). A Prospective Observational Study of Long-term Outcomes.
Brief Title: Guided Optimisation of Long-term Disease rEduction in secoNdary Prevention of CVD
Acronym: GOLDEN
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Network for Cardiovascular Research (WCN), Utrecht (Unknown); Novartis Pharmaceuticals (Industry); Amarin Pharma Inc. (Industry)
Responsible Party: Principal Investigator, Harald Jorstad, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2023.0331
Record Dates: First submitted 2024-07-05; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Acute Coronary Syndrome
Keywords: Cardiovascular prevention; Coronary revascularisation; Pharmacological approach; Teachable moment; Major cardiovascular events; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 'Current practice' group: The 'current practice' treated patients' group will provide data on current practices in the preventive treatment after hospitalization for acute coronary syndrome or coronary revascularization. (i.e. incremental, individual titration at treating physician's discretion)
  Interventions: Other: No intervention (observational study)
- 'First-time-right' (FTR) group: In line with the 2021 ESC Prevention guidelines, the FTR group will be treated according to the 'first-time-right' strategy(1). While no specific therapeutic protocols are mandated by our observational study, participating centers will be required to apply the 'first-time- right' strategy: i.e. the direct, in-hospital initiation or planned initiation of all guideline-recommended preventive pharmacotherapeutic treatments.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention, only guideline implementation (observational study)

SUMMARY:
The goal of this observational study is to evaluate the implementation of a 'first-time-right' pharmacological treatment strategy in patients hospitalized with coronary artery disease.

The main question it aims to answer is:

Does early (immediately post-event) initiation of a full set of guideline-based, individualized, preventive medication lead to reductions in cardiovascular events compared to current practice (incremental titration strategies)?

Researchers will compare the 'first-time-right' strategy group to the current practice group to see if there are improvements in major adverse cardiac and cerebrovascular events (MACE) at 36 months.

Participants will:

* Receive either the 'first-time-right' strategy or current practice for secondary prevention.
* Be monitored (data collection) through routine clinical visits at baseline, 8 weeks, 12, and additional telephone contacts at 24, and 36 months after discharge.
* Complete online questionnaires at hospitalization, 8 weeks, 12, 24, and 36 months after discharge.

DETAILED DESCRIPTION:
Rationale:

Individuals with clinically established coronary artery disease are at high risk of recurrent events and death. To reduce this risk, incremental titration of preventive medication to reach pre-defined risk factor targets is recommended by international guidelines.

However, using this approach, disappointing reductions in risk are generally attained, mainly resulting from inadequate use of preventive medication. The European 2021 Prevention guidelines recommend compressing preventive strategies into a maximum of two steps: first, attainment of 'minimal' risk-factor targets, followed by rapid individualized residual risk management (1). While the conventional interpretation of preventive guidelines has led to medication titration over months or even years, - with suboptimal results, the new guideline-based approach de facto constitutes a front-loaded, 'first- time-right' strategy, where as early as during hospitalization, a complete medication plan is formulated and implemented. However, the practical implementation and effects on clinical outcomes of such a strategy have not been investigated. The investigators therefore aim to investigate the effects of implementing a 'first-time-right' guideline-based pharmacological treatment strategy, compared to current incremental, individual-titration strategies, in patients hospitalized with coronary artery disease. As both treatment strategies constitute a different application of current international guidelines, no experimental treatments are included. The investigators will therefore conduct an observational study to investigate the effects of both strategies. The investigators hypothesize that application of the first-time-right pharmacological strategy, i.e. early (immediately post-event) initiation of a full set of guideline-based, individualized, preventive medications will lead to greater risk factor control, and to reductions in cardiovascular events, compared to current practice (i.e. incremental titration strategies).

Goals:

Primary Objective: To evaluate the impact of a 'first-time-right' pharmacological risk factor management strategy, according to the European 2021 Prevention guidelines, compared with current practice (i.e. incremental titration) on major adverse cardiac- and cerebrovascular events (MACE, 4-point: CVD death, myocardial infarction, (ischemic or hemorrhagic) stroke, and ischemia-driven revascularization) at 36 months. Secondary objectives: CVD death, myocardial infarction, stroke, and ischemia-driven revascularization (plus in 2 and 3-point MACE combinations), acute limb ischemia, carotid revascularization, unplanned cardiovascular hospital readmission, improvement in cardiovascular risk factors (drug- targeted and lifestyle-related risk factors), self-reported medication use and adherence scores, quality of life.

Study design:

GOLDEN is a prospective, observational study designed to evaluate the implementation of the guideline-based 'first-time-right' strategy in at least 30 cardiology departments in the Netherlands (Figure 1, Appendix). Study supervision, including data management and statistical analyses of the study, will be performed and coordinated at the Amsterdam UMC, assisted by the Dutch Network forCardiovascular Research (WCN), Utrecht, The Netherlands.

The study will be embedded in the collaboration of the partners of the Dutch Cardiovascular Alliance, supporting the goal of reducing the cardiovascular disease burden in The Netherlands by collaboration in research and implementation. Amsterdam UMC has the role of sponsor and is responsible for the scientific and operational leadership. When all relevant national partners support the implementation goal of First Time Right, participating centers will be recruited within the academic centers (through NetherLands Heart Institute, NLHI) and non-academic centers (through the Dutch Network for Cardiovascular Research, WCN), Utrecht, The Netherlands. Patient data will be captured and stored in an electronic database (Castor) and will only be available for the investigator (sponsor). WCN (Werkgroep Cardiologische centra Nederland) is a research network of cardiovascular investigators (www.WCN.life). The network consists of nearly 60 cardiovascular research departments across the Netherlands. The WCN office provides central support to both the sponsor and the participating sites through central feasibility, site ID, contracting, recruitment and quality support. The research professionals are employed by each individual site. Data on patient inclusion and data quality will be shared with WCN for quality assurance purposes. No individual patient data will be shared with WCN.

Our observational study comprises two groups:1) The 'current practice' group, constituting current secondary prevention practices treated patients (i.e. incremental, individual titration at treating physician's discretion) 2) The 'first-time-right' group, when the 'first- time-right' guideline-based strategy is implemented. The study program is outlined in Figure 2 (Appendix). All centers will start including in the 'current practice' arm. After inclusion of 50% of the sample size, a blanking period of 8 weeks will be observed, where no inclusions will take place in any center. This time period will be used to train all participating centers in the 'first-time-right' strategy.

Subsequently, all centers will proceed to include in the 'first-time- right' cohort. The 'current practice' treated patients' group will provide data on current practices in the preventive treatment after hospitalization for acute coronary syndrome or coronary revascularization.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age (no upper limit)
* Coronary event, i.e. ACS or coronary revascularisation
* Able to provide informed consent

Exclusion Criteria:

* (short-term planned) pregnancy or breast feeding
* Dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all patients who have consented to the use of their clinical data and who are hospitalized at cardiology departments of participating hospitals (Dutch Network for Cardiovascular Research (WCN and University Medical Centers) in the Netherlands.
Sampling Method: Probability Sample
Enrollment: 5586 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
4-point MACE | 36 months
  Composite of cardiovascular death, myocardial infarction, any documented stroke (ischemic or hemorrhagic), ischemia-driven revascularization.

SECONDARY OUTCOMES:
Uncombined MACE evaluations | 8 weeks, 12 months, 24 months, 36 months after discharge
  Cardiovascular death, myocardial infarction, (ischemic or hemorrhagic) stroke, ischemia-driven revascularization (uncombined evaluation)
Combined outcomes: 2-point and 3-point MACE | 8 weeks, 12 months, 24 months, 36 months after discharge
  Combined outcomes:
  2-point MACE: CVD death, MI, and 3-point MACE: CVD death, MI, revascularization
Extended MACE | 8 weeks, 12 months, 24 months, 36 months after discharge
  4-point MACE, in addition to two additional arterial atherosclerotic outcomes: acute limb ischemia and carotid revascularization 2-point MACE: CVD death, MI, and 3-point MACE: CVD death, MI, revascularization
Unplanned cardiovascular hospital readmission | 8 weeks, 12 months, 24 months, 36 months after discharge
  Unplanned cardiovascular hospital readmission
LDL-cholesterol | baseline= (max. 3 months) prior to event or revascularisation procedure, 8 weeks, 12 months after discharge
  mmol/L
Diastolic blood pressure | baseline= (max. 3 months) prior to event or revascularisation procedure, 8 weeks, 12 months after discharge
  mmHg
C-reactive protein | baseline= (max. 3 months) prior to event or revascularisation procedure, 8 weeks, 12 months after discharge
  mg/L
Fasting glucose | baseline= (max. 3 months) prior to event or revascularisation procedure, 8 weeks, 12 months after discharge
  mmol/L
HbA1c | baseline= (max. 3 months) prior to event or revascularisation procedure, 8 weeks, 12 months after discharge
  mmol/mol
Systolic blood pressure | baseline= (max. 3 months) prior to event or revascularisation procedure, 8 weeks, 12 months after discharge
  mmHg
Medication Adherence Report Scale (MARS5) | baseline= between event or coronary intervention and discharge, 8 weeks, 12 months, 24 months, 36 months
  5 questions about medication adherence (Horne et al. 2005, Chan et al. 2020)
visual analog scale (VAS) medication adherence | baseline= between event or coronary intervention and discharge, 8 weeks, 8 weeks, 12 months, 24 months, 36 months
  Scale 0-100%. Hihger score indicating better medication adherence
Beliefs about Medicine (BMQ) | baseline= between event or coronary intervention and discharge, 8 weeks, 8 weeks, 12 months, 24 months, 36 months
  BMQ: Beliefs about medicine questionnaire -specific part only (Horne et al. 1999) Questionnaire (BMQ)
Quality-of-Life (QoL) | baseline= between event or coronary intervention and discharge, 8 weeks, 8 weeks, 12 months, 24 months, 36 months
  EuroQoL-5D questionnaire (EuroQol group, 1990) Questionnaire (BMQ)

OTHER OUTCOMES:
The iMTA Medical Consumption Questionnaire (iMCQ) | baseline= between event or coronary intervention and discharge, 8 weeks, 12 months, 36 months
  measuring medical consumption
The iMTA Productivity Cost Questionnaire | baseline= between event or coronary intervention and discharge, 8 weeks, 12 months, 36 months
  measuring productivity cost

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein Snaterse, dr., Study Chair — Amsterdam UMC; Fabrice M.A.C. Martens, Prof. dr., Study Chair — Amsterdam UMC; Harald T. Jorstad, dr., Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Angelantonio ED, Franco OH, Halvorsen S, Richard Hobbs FD, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice: Developed by the Task Force for cardiovascular disease prevention in clinical practice with representatives of the European Society of Cardiology and 12 medical societies With the special contribution of the European Association of Preventive Cardiology (EAPC). Rev Esp Cardiol (Engl Ed). 2022 May;75(5):429. doi: 10.1016/j.rec.2022.04.003. No abstract available. English, Spanish. PMID 35525570